CLINICAL TRIAL: NCT01767194
Title: A Phase II Randomized Trial of Irinotecan/Temozolomide With Temsirolimus (NSC# 683864) or Chimeric 14.18 Antibody (Ch14.18) (NSC# 764038) in Children With Refractory, Relapsed or Progressive Neuroblastoma
Brief Title: Irinotecan Hydrochloride and Temozolomide With Temsirolimus or Dinutuximab in Treating Younger Patients With Refractory or Relapsed Neuroblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03125; NCI-2012-03125 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000745188; ANBL1221; COG-ANBL1221; PANBL1221_A08PAMDREVW01; ANBL1221 (Other: Children's Oncology Group); ANBL1221 (Other: CTEP); U10CA180886 (NIH); U10CA098543 (NIH)
Record Dates: First submitted 2013-01-09; First posted 2013-01-14 (Estimated); Results first posted 2019-11-18 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Ganglioneuroblastoma; Recurrent Neuroblastoma
MeSH Terms: conditions — Ganglioneuroblastoma; Neuroblastoma | interventions — dinutuximab; Irinotecan; sargramostim; Colony-Stimulating Factors; Temozolomide; temsirolimus; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (temozolomide, irinotecan hydrochloride, temsirolimus) (Experimental): CLOSED TO ACCRUAL 06/17/2016 Patients receive temozolomide PO on days 1-5, irinotecan hydrochloride IV over 90 minutes on days 1-5, and temsirolimus IV over 30 minutes on days 1 and 8.
  Interventions: Drug: Irinotecan Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Temozolomide; Drug: Temsirolimus
- Arm II (temozolomide, irinotecan hydrochloride, dinutuximab) (Experimental): Patients receive temozolomide PO on days 1-5, irinotecan hydrochloride over 90 minutes on days 1-5, dinutuximab IV over 10-20 hours on days 2-5, and sargramostim SC or IV over 2 hours on days 6-12.
  Interventions: Biological: Dinutuximab; Drug: Irinotecan Hydrochloride; Other: Laboratory Biomarker Analysis; Biological: Sargramostim; Drug: Temozolomide

INTERVENTIONS:
Biological: Dinutuximab — Given IV
  Other Names: Ch 14.18UTC; Ch14.18; MOAB Ch14.18; monoclonal antibody Ch14.18; Unituxin
  Arms: Arm II (temozolomide, irinotecan hydrochloride, dinutuximab)
Drug: Irinotecan Hydrochloride — Given IV
  Other Names: Campto; Camptosar; Camptothecin 11; Camptothecin-11; CPT 11; CPT-11; Irinomedac; Irinotecan Hydrochloride Trihydrate; Irinotecan Monohydrochloride Trihydrate; U-101440E
Other: Laboratory Biomarker Analysis — Optional correlative studies
Biological: Sargramostim — Given SC or IV
  Other Names: 23-L-Leucinecolony-Stimulating Factor 2; DRG-0012; Leukine; Prokine; rhu GM-CFS; Sagramostim; Sargramostatin
  Arms: Arm II (temozolomide, irinotecan hydrochloride, dinutuximab)
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temodal; Temodar; Temomedac; TMZ
Drug: Temsirolimus — Given IV
  Other Names: CCI-779; CCI-779 Rapamycin Analog; Cell Cycle Inhibitor 779; Rapamycin Analog; Rapamycin Analog CCI-779; Torisel
  Arms: Arm I (temozolomide, irinotecan hydrochloride, temsirolimus)

SUMMARY:
This randomized phase II trial studies how well irinotecan hydrochloride and temozolomide with temsirolimus or dinutuximab work in treating younger patients with neuroblastoma that has returned or does not respond to treatment. Drugs used in chemotherapy, such as irinotecan hydrochloride and temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Temsirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as dinutuximab, may find tumor cells and help kill them or carry tumor-killing substances to them. It is not yet known whether giving irinotecan hydrochloride and temozolomide together with temsirolimus or dinutuximab is more effective in treating neuroblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify whether temsirolimus or ch14.18 (dinutuximab) is the optimal therapeutic agent to consider for further testing in a future Phase III randomized trial for treatment of newly diagnosed high-risk neuroblastoma.

II. To determine the response rate of patients with relapsed, refractory or progressive neuroblastoma following treatment with irinotecan, temozolomide and ch14.18 (dinutuximab) and to compare this with the known response rate of patients treated with irinotecan and temozolomide alone.

EXPLORATORY OBJECTIVES:

I. To compare the response rates (RR) for patients receiving temsirolimus or ch14.18 (dinutuximab) in combination with irinotecan (irinotecan hydrochloride) and temozolomide.

II. To compare the progression free survival (PFS) and overall survival (OS) rates for patients receiving temsirolimus or ch14.18 (dinutuximab) in combination with irinotecan and temozolomide.

III. To compare the toxicities associated with temsirolimus or ch14.18 (dinutuximab) when combined with irinotecan and temozolomide in patients with refractory, relapsed or progressive neuroblastoma.

IV. To compare the ability to maintain intended dose intensity of all agents when temsirolimus or ch14.18 (dinutuximab) is combined with irinotecan and temozolomide in patients with refractory, relapsed or progressive neuroblastoma.

V. To determine the concordance between tumor responses as defined by standard International Neuroblastoma Response Criteria (INRC) versus response per the revised INRC.

VI. To study the clinical relevance of naturally occurring anti-glycan antibodies in patients receiving ch14.18 (dinutuximab) antibody.

VII. To study the clinical relevance of natural killer (NK) receptor natural cytotoxicity triggering receptor 3 (NKp30) isoforms in patients receiving ch14.18 (dinutuximab) antibody or temsirolimus.

VIII. To study the association between host factors and response to irinotecan, temozolomide and ch14.18 (dinutuximab).

IX. To characterize the tumor immune-microenvironment (gene expression; immune effector cells, activities and signaling molecules; immune target expression) following treatment with irinotecan, temozolomide and ch14.18 (dinutuximab).

X. To study the association between changes in the tumor immune-microenvironment (gene expression; immune effector cells, activities and signaling molecules; immune target expression) with response following treatment with irinotecan, temozolomide and ch14.18 (dinutuximab).

XI. To study the association between tumor genomic and transcriptomic aberrations as well as levels of circulating ganglioside (GD2) with response to irinotecan, temozolomide and ch14.18 (dinutuximab).

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I (CLOSED TO ACCRUAL 06/17/2016): Patients receive temozolomide orally (PO) on days 1-5, irinotecan hydrochloride intravenously (IV) over 90 minutes on days 1-5, and temsirolimus IV over 30 minutes on days 1 and 8.

ARM II: Patients receive temozolomide PO on days 1-5, irinotecan hydrochloride over 90 minutes on days 1-5, dinutuximab IV over 10-20 hours on days 2-5, and sargramostim subcutaneously (SC) or IV over 2 hours on days 6-12.

In both arms, treatment repeats every 21 days for up to 17 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have had histologic verification of neuroblastoma or ganglioneuroblastoma or demonstration of neuroblastoma cells in the bone marrow with elevated urinary catecholamines (i.e., > 2 x upper limit of normal [ULN]), at the time of initial diagnosis
* For the purposes of this study, aggressive multidrug chemotherapy is defined as chemotherapy including 2 or more agents that must include an alkylating agent and a platinum-containing compound; patients must have ONE of the following:

  * First episode of recurrent disease following completion of aggressive multi-drug frontline therapy
  * First episode of progressive disease during aggressive multi-drug frontline therapy
  * Primary resistant/refractory disease (less than partial response by INRC) detected at the conclusion of at least 4 cycles of aggressive multidrug induction chemotherapy on or according to a high-risk neuroblastoma protocol (examples include A3973, ANBL0532, ANBL09P1, etc.)
* Patients must have at least ONE of the following:

  * Measurable tumor on magnetic resonance imaging (MRI), computed tomography (CT) scan obtained within 3 weeks prior to study entry; measurable is defined as >= 10 mm in at least one dimension on spiral/helical CT that is metaiodobenzylguanidine (MIBG) avid or demonstrates increased fludeoxyglucose (FDG) uptake on positron emission tomography (PET) scan
  * MIBG scan obtained within 3 weeks prior to study entry with positive uptake at a minimum of one site; this site must represent disease recurrence after completion of therapy, progressive disease on therapy, or refractory disease during induction
  * Patients with resistant/refractory soft tissue disease that is not MIBG avid or does not demonstrate increased FDG uptake on PET scan must undergo biopsy to document the presence of viable neuroblastoma; biopsy is not required for patients who have new site of soft tissue disease (radiographic evidence of disease progression) regardless of whether progression occurs while receiving therapy or after completion of therapy
  * Note: Patients with elevated catecholamines (i.e., > 2 x ULN) only or bone marrow disease only are NOT eligible for this study
* Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0, 1 or 2; use Karnofsky for patients > 16 years of age and Lansky for patients =< 16 years of age
* Patients must have received frontline therapy (including surgery, chemotherapy, autologous stem cell transplant [SCT] +/- MIBG, immunotherapy, radiotherapy, and retinoids) but may NOT have received second line chemotherapy for resistant/refractory, relapsed disease or progressive disease
* At least 14 days must have elapsed since completion of myelosuppressive therapy
* At least 7 days must have elapsed since the completion of therapy with a non-myelosuppressive biologic agent or retinoid
* No interim time prior to study entry is required following prior radiation therapy (RT) for non-target lesions; however, patients must not have received radiation for a minimum of 4 weeks prior to study entry at the site of any lesion that will be identified as a target lesion to measure tumor response; lesions that have been previously radiated cannot be used as target lesions unless there is radiographic evidence of progression at the site following radiation or a biopsy done following radiation shows viable neuroblastoma; palliative radiation is allowed to sites that will not be used to measure response during this study
* Patients are eligible >= 6 weeks after autologous stem cell transplants or stem cell infusions as long as hematologic and other eligibility criteria have been met
* Patients are eligible >= 6 weeks after therapeutic 131I-MIBG provided that all other eligibility criteria are met
* Subjects who have previously received anti-GD2 monoclonal antibodies for biologic therapy or for tumor imaging are eligible unless they have had progressive disease while receiving prior anti-GD2 therapy; subjects who have received autologous marrow infusions or autologous stem cell infusions that were purged using monoclonal antibody linked to beads, but no other form of anti-GD2 monoclonal antibody, are eligible
* Patients must not have received long-acting myeloid growth factors (e.g., Neulasta) within 14 days of entry on this study; seven days must have elapsed since administration of a short acting myeloid growth factor
* Peripheral absolute neutrophil count (ANC) >= 750/uL
* Platelet count >= 75,000/uL (transfusion independent)
* Patients known to have bone marrow involvement with neuroblastoma are eligible provided that minimum ANC and platelet count criteria are met but are not evaluable for hematological toxicity
* Creatinine clearance or estimated radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 or
* A serum creatinine =< upper limit of normal (ULN) based on age/gender as follows:

  * Age 1 month to < 6 months: 0.4 for males, 0.4 for females
  * Age 6 months to < 1 year: 0.5 for males, 0.5 for females
  * Age 1 to < 2 years: 0.6 for males, 0.6 for females
  * Age 2 to < 6 years: 0.8 for males, 0.8 for females
  * Age 6 to < 10 years: 1 for males, 1 for females
  * Age 10 to < 13 years: 1.2 for males, 1.2 for females
  * Age 13 to < 16 years: 1.5 for males, 1.4 for females
  * Age >= 16 years: 1.7 for males, 1.4 for females
* Total bilirubin =< 1.5 x ULN for age AND
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 5.0 x ULN for age (=< 225 U/L); for the purpose of this study, the ULN for SGPT is 45 U/L
* Adequate central nervous system function defined as:

  * Patients with a history of central nervous system (CNS) disease must have no clinical or radiological evidence of CNS disease at the time of study enrollment
  * Patients with seizure disorders may be enrolled if seizures are well controlled on anticonvulsants
  * CNS toxicity =< grade 2
* Shortening fraction of >= 27% by echocardiogram (ECHO) OR
* Ejection fraction >= 50% by ECHO or gated radionuclide study
* Adequate coagulation defined as:

  * Prothrombin time (PT) =< 1.2 x upper limit of normal
* Adequate pulmonary function defined as:

  * No evidence of dyspnea at rest, no exercise intolerance, no chronic oxygen requirement, and room air pulse oximetry > 94% if there is a clinical indication for pulse oximetry; normal pulmonary function tests in patients who are capable of cooperating with testing (including diffusion capacity of the lung of carbon monoxide [DLCO]) are required if there is a clinical indication for determination; for patients who do not have respiratory symptoms, full pulmonary function tests (PFTs) are NOT required

Exclusion Criteria:

* Men and women of childbearing potential and their partners must agree to use adequate contraception while enrolled on this study; based on the established teratogenic potential of alkylating agents, pregnant women will be excluded from this study; female patients who are lactating must agree to stop breastfeeding or will otherwise be excluded from this study; females of childbearing potential must have a negative pregnancy test to be eligible for this study
* Patients with elevated catecholamines (i.e., > 2 x ULN) only or bone marrow disease only are NOT eligible for this study
* Patients must have been off pharmacologic doses of systemic steroids for at least 7 days prior to enrollment; patients who require or are likely to require pharmacologic doses of systemic corticosteroids while receiving treatment on this study are ineligible; the only exception is for patients known to require 2 mg/kg or less of hydrocortisone (or an equivalent dose of an alternative corticosteroid) as premedication for blood product administration in order to avoid allergic transfusion reactions; the use of conventional doses of inhaled steroids for the treatment of asthma is permitted, as is the use of physiologic doses of steroids for patients with known adrenal insufficiency
* Patients must not have received enzyme-inducing anticonvulsants including phenytoin, phenobarbital, valproic acid, or carbamazepine for at least 7 days prior to study enrollment; patients receiving non-enzyme inducing anticonvulsants such as gabapentin or levetiracetam will be eligible
* Patients must not have been diagnosed with myelodysplastic syndrome or with any malignancy other than neuroblastoma
* Patients with symptoms of congestive heart failure are not eligible
* Patients must not have >= grade 2 diarrhea
* Patients must not have uncontrolled infection
* Patients with a history of grade 4 allergic reactions to anti-GD2 antibodies or reactions that required discontinuation of the anti-GD2 therapy are not eligible
* Patients with a significant intercurrent illness (any ongoing serious medical problem unrelated to cancer or its treatment) that is not covered by the detailed exclusion criteria and that is expected to interfere with the action of study agents or to significantly increase the severity of the toxicities experienced from study treatment are not eligible

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2013-02-12 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajen Mody, Principal Investigator — Children's Oncology Group
Locations (157):
- United States (136):
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lee Memorial Health System, Fort Myers, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Winthrop Hospital, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (5):
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Children's Hospital-Brisbane, Herston, Queensland
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (13):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec
- New Zealand (2):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch
- San Jorge Children's Hospital, San Juan, Puerto Rico

REFERENCES:
- [Derived] Erbe AK, Diccianni MB, Mody R, Naranjo A, Zhang FF, Birstler J, Kim K, Feils AS, Hung JT, London WB, Shulkin BL, Mathew V, Parisi MT, Servaes S, Asgharzadeh S, Maris JM, Park J, Yu AL, Sondel PM, Bagatell R. KIR/KIR-ligand genotypes and clinical outcomes following chemoimmunotherapy in patients with relapsed or refractory neuroblastoma: a report from the Children's Oncology Group. J Immunother Cancer. 2023 Feb;11(2):e006530. doi: 10.1136/jitc-2022-006530. PMID 36822669
- [Derived] Mody R, Yu AL, Naranjo A, Zhang FF, London WB, Shulkin BL, Parisi MT, Servaes SE, Diccianni MB, Hank JA, Felder M, Birstler J, Sondel PM, Asgharzadeh S, Glade-Bender J, Katzenstein H, Maris JM, Park JR, Bagatell R. Irinotecan, Temozolomide, and Dinutuximab With GM-CSF in Children With Refractory or Relapsed Neuroblastoma: A Report From the Children's Oncology Group. J Clin Oncol. 2020 Jul 1;38(19):2160-2169. doi: 10.1200/JCO.20.00203. Epub 2020 Apr 28. PMID 32343642
- [Derived] Mody R, Naranjo A, Van Ryn C, Yu AL, London WB, Shulkin BL, Parisi MT, Servaes SE, Diccianni MB, Sondel PM, Bender JG, Maris JM, Park JR, Bagatell R. Irinotecan-temozolomide with temsirolimus or dinutuximab in children with refractory or relapsed neuroblastoma (COG ANBL1221): an open-label, randomised, phase 2 trial. Lancet Oncol. 2017 Jul;18(7):946-957. doi: 10.1016/S1470-2045(17)30355-8. Epub 2017 May 23. PMID 28549783

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Temozolomide, Irinotecan Hydrochloride, Temsirolimus) | Arm II (Temozolomide, Irinotecan Hydrochloride, Dinutuximab)
Started | 19 | 54
Completed | 1 | 11
Not Completed | 18 | 43
Not completed — Adverse Event | 1 | 1
Not completed — Death | 0 | 1
Not completed — Lack of Efficacy | 12 | 11
Not completed — Physician Decision | 2 | 23
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Ineligible | 1 | 1
Not completed — Refusal by patient/parent | 2 | 4
Not completed — Criteria not met on time for next cycle | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Temozolomide, Irinotecan Hydrochloride, Temsirolimus) | Arm II (Temozolomide, Irinotecan Hydrochloride, Dinutuximab) | Total
Number analyzed (Participants) | 19 | 54 | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19 | 54 | 73
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: Years] | 7.2 [2.9 to 16.2] | 4.9 [1.3 to 15.9] | 5.7 [1.3 to 16.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 21 | 29
  Male | 11 | 33 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 8 | 13
  Not Hispanic or Latino | 14 | 43 | 57
  Unknown or Not Reported | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 3 | 7 | 10
  White | 14 | 36 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 6 | 7
Region of Enrollment [Number; unit: participants]
  United States | 15 | 45 | 60
  Canada | 2 | 5 | 7
  Australia | 2 | 2 | 4
  New Zealand | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Randomized Patients Who Are Responders
Description: The percentage of patients who are responders will be tabulated, including a 95% confidence interval on the response rate. Responders are defined as patients who achieve a best overall response of complete response (CR), very good partial response (VGPR), or partial response (PR) per the International Neuroblastoma Response Criteria (INRC). Per INRC: CR= Disappearance of all target lesions. No evidence of tumor at any site; VGPR= >90% decrease of the disease measurement for CT/MRI target lesions. All pre-existing bone lesions with CR by MIBG; MIBG scan can be stable disease (SD) or CR in soft tissue lesions corresponding to lesions on CT/MRI. CR in bone marrow. No new sites of tumor; PR= >=30% decrease in the disease measurement for CT/MRI target lesions. Bone marrow with CR. MIBG with either PR/CR in bone lesions; MIBG may be SD or CR in soft tissue lesions corresponding to lesions on CT/MRI. Homovanillic acid (HVA)/Vanillylmandelic acid (VMA) may still be elevated.
Time Frame: Up to the first 6 cycles of treatment
Population: Includes all eligible patients randomly assigned to Arm I or Arm II. Of the 19 participants randomized to Arm I, one was ineligible and not included in the analysis. Of the 54 participants assigned to Arm II, 1 was ineligible and 36 were non-randomly assigned, and not included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Arm I (Temozolomide, Irinotecan Hydrochloride, Temsirolimus) | Arm II (Temozolomide, Irinotecan Hydrochloride, Dinutuximab)
Number analyzed (Participants) | 18 | 17
Percentage of patients | 5.6 [0.0 to 16.1] | 52.9 [29.2 to 76.7]

2. Primary Outcome: Percentage of Patients in the Dinutuximab Arm Who Are Responders
Description: Percentage of patients who are responders to therapy with dinutuximab will be tabulated, including a 95% confidence interval on the response rate. Responders are defined as patients who achieve a best overall response of complete response (CR), very good partial response (VGPR), or partial response (PR) per the International Neuroblastoma Response Criteria (INRC). Per INRC: CR= Disappearance of all target lesions. No evidence of tumor at any site; VGPR= >90% decrease of disease measurement for CT/MRI target lesions. All pre-existing bone lesions with CR by MIBG; MIBG scan can be stable disease (SD) or CR in soft tissue lesions corresponding to lesions on CT/MRI. CR in bone marrow. No new sites of tumor; PR= ≥30% decrease in disease measurement for CT/MRI target lesions. Bone marrow with CR. MIBG with either PR/CR in bone lesions; MIBG may be SD or CR in soft tissue lesions corresponding to lesions on CT/MRI. Homovanillic acid (HVA)/ Vanillylmandelic acid (VMA) may still be elevated.
Time Frame: Up to the first 6 cycles of treatment
Population: Includes all eligible patients either randomized or non-randomly assigned to Arm II. Of the 54 participants assigned to Arm II, 1 was ineligible and not included in the analysis. The remaining 53 eligible participants are included in the analysis, 17 randomized and 36 non-randomly assigned to Arm II.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Arm II (Temozolomide, Irinotecan Hydrochloride, Dinutuximab)
Number analyzed (Participants) | 53
Percentage of patients | 41.2 [28.2 to 54.8]

3. Other Pre Specified Outcome: Progression-free Survival
Description: Kaplan-Meier method will be used to estimate progression-free survival. Progression-free survival will be defined as the time from enrollment to relapse, progressive disease, or death attributable to tumor or treatment.
Time Frame: Up to 3 years
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Overall Survival
Description: Kaplan-Meier method will be used to estimate overall survival. Overall survival is defined as the time from enrollment on the study until death.
Time Frame: Up to 3 years
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Occurrence of Unacceptable Toxicities
Description: The proportion of patients with at least one grade 3 or higher toxicity, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0.
Time Frame: Up to 1 year
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Ability to Maintain Intended Treatment Without a Dose Reduction or Going Off Protocol Therapy for Toxicity
Description: The proportion of patients who required a dose modification or went off protocol therapy for toxicity will be calculated for each treatment group.
Time Frame: Up to 1 year
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Overall Response
Description: The proportion of patients achieving each type of overall response (complete response, partial response, stable disease, progressive disease) will be calculated according to the International Neuroblastoma Response Criteria (INRC).
Time Frame: Up to the first 6 cycles of treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Through completion of protocol therapy, up to approximately 1 year.
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution, via expedited reporting (NCI AdEERs / CAeRs). The "AE Other" table reflects all CTCAEs collected excluding those that were reported as SAEs. Ineligible patients and patients that reported not receiving treatment are excluded from reporting of adverse events.
Arm/Group | Arm I (Temozolomide, Irinotecan Hydrochloride, Temsirolimus) | Arm II (Temozolomide, Irinotecan Hydrochloride, Dinutuximab)
All-Cause Mortality (participants affected / at risk) | 12/18 | 15/51
Serious Adverse Events (participants affected / at risk) | 5/18 | 18/51
Other Adverse Events (participants affected / at risk) | 10/18 | 39/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Temozolomide, Irinotecan Hydrochloride, Temsirolimus) (N=18) | Arm II (Temozolomide, Irinotecan Hydrochloride, Dinutuximab) (N=51)
Alanine aminotransferase increased (Investigations) | 1 | 1
Allergic reaction (Immune system disorders) | 1 | 0
Anaphylaxis (Immune system disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 2
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 2
BACTEREMIA - LINE INFECTIONS (Infections and infestations) | 0 | 1
BLOOD (Infections and infestations) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Creatinine increased (Investigations) | 0 | 1
Death NOS (General disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Fever (General disorders) | 1 | 1
GGT increased (Investigations) | 1 | 1
Headache (Nervous system disorders) | 0 | 1
Hearing impaired (Ear and labyrinth disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Mucosal infection (Infections and infestations) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 4
norovirus (Infections and infestations) | 0 | 1
Pain (General disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Platelet count decreased (Investigations) | 1 | 0
POSITIVE BLOOD CULTURES (Infections and infestations) | 1 | 0
Prolapse of intestinal stoma (Injury, poisoning and procedural complications) | 0 | 1
RSV (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Small intestine infection (Infections and infestations) | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 1
TEMPORARY VISION LOSS (Eye disorders) | 0 | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Upper respiratory infection (Infections and infestations) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Urine output decreased (Investigations) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Weight loss (Investigations) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2
White blood cell decreased (Investigations) | 2 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Temozolomide, Irinotecan Hydrochloride, Temsirolimus) (N=18) | Arm II (Temozolomide, Irinotecan Hydrochloride, Dinutuximab) (N=51)
Abdominal pain (Gastrointestinal disorders) | 0 | 3
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 4 | 8
Allergic reaction (Immune system disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 5 | 12
Anorexia (Metabolism and nutrition disorders) | 2 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
BACTEREMIA (Infections and infestations) | 0 | 1
BLOOD (Infections and infestations) | 1 | 0
BLOOD - STAPHYLOCOCCUS EPIDERMIDIS ISOLATED. (Infections and infestations) | 0 | 1
BLOOD - STAPHYLOCOCCUS HOMINIS ISOLATES (Infections and infestations) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Blurred vision (Eye disorders) | 0 | 1
Capillary leak syndrome (Vascular disorders) | 0 | 2
Cardiac arrest (Cardiac disorders) | 0 | 1
CENTRAL LINE INFECTION (Infections and infestations) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 3
Delirium (Psychiatric disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 1
Fatigue (General disorders) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Fever (General disorders) | 0 | 10
GGT increased (Investigations) | 0 | 2
GRAM-POSITIVE BACILLI FROM PORT BLOOD CULTURE (Infections and infestations) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 3
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 4
Hypokalemia (Metabolism and nutrition disorders) | 4 | 9
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 1
Hypotension (Vascular disorders) | 0 | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 4
INFECTION (Infections and infestations) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Irritability (Psychiatric disorders) | 0 | 2
LINE INFECTION (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Lymphocyte count decreased (Investigations) | 4 | 13
Lymphocyte count increased (Investigations) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Neutrophil count decreased (Investigations) | 7 | 13
Non-cardiac chest pain (General disorders) | 0 | 1
Oral pain (Gastrointestinal disorders) | 1 | 0
Pain (General disorders) | 0 | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Platelet count decreased (Investigations) | 5 | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
RESPIRATORY SYNCTIAL VIRUS (RSV) FROM NASAL SWAB (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 1 | 1
STAPH. WARNERI FROM WHITE LUMEN (Infections and infestations) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 3
Urine output decreased (Investigations) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 5
Weight gain (Investigations) | 0 | 1
White blood cell decreased (Investigations) | 4 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-19): https://cdn.clinicaltrials.gov/large-docs/94/NCT01767194/Prot_SAP_000.pdf